CLINICAL TRIAL: NCT01386164
Title: Immune Response to Bivalent and Tetravalent Human Papillomavirus Vaccine in HIV Infected Adults
Acronym: HIPAVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTN0001
Record Dates: First submitted 2011-06-22; First posted 2011-06-30 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: HIV; Human Papillomavirus
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gardasil® (Experimental)
  Interventions: Biological: Gardasil
- Cervarix® (Experimental)
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Gardasil — Subjects will receive three doses of the study vaccine administered intramuscularly according to a Day 0, Week 6, and Month 6 vaccination schedule.
  Other Names: Tetravalent HPV vaccine
  Arms: Gardasil®
Biological: Cervarix — Subjects will receive three doses of the study vaccine administered intramuscularly according to a Day 0, Week 6, and Month 6 vaccination schedule.
  Other Names: Bivalent HPV vaccine
  Arms: Cervarix®

SUMMARY:
The purpose of this study is to analyze and compare the immunogenicity of Bivalent and Tetravalent vaccines against Human Papillomavirus in HIV-infected adult persons.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive subjects.
* Age above 18 at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Subjects whom the investigator believes can and will comply with the requirements of the protocol.
* If currently on antiretroviral therapy (ART), subjects must be compliant to triple therapy (highly active ART) and have undetectable viral load for a period of six months prior to study entry.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject has a negative pregnancy test at screening and on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period.

Exclusion Criteria:

* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (Day 0 to Month 12).
* Pregnant or breastfeeding female.
* Previous enrollment in the study.
* Subjects whom the investigator believes cannot and/or will not comply with the requirements of the protocol (i.e. because of abuse of drugs or alcohol, dementia or given medical, psychiatric, social or work related conditions).
* Chronic administration of immunosuppressive drugs
* Cancer or autoimmune disease
* Previous allergic reaction to vaccination
* Known allergy towards on or more components of either of the test drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Geometric mean titres of serum HPV-16 and HPV-18 antibody titers on measured by Pseudovirion-Based Neutralization Assay (PBNA) | Day 0, Day 45, Day 180, Day 210 and Day 365

SECONDARY OUTCOMES:
Geometric mean titres of serum HPV-31, HPV-33, HPV-45, HPV-52 and HPV-58 antibody measured by Pseudovirion-Based Neutralization Assay (PBNA) | Day 0, Day 45, Day 180, Day 210 and Day 365
Avidity of HPV-16 and -18 serum antibodies measured by ELISA | Day 0, Day 45, Day 180, Day 210 and Day 365
Frequencies of HPV-16 and HPV-18 T-cells measured by flow cytometry | Day 0, Day 45, Day 180, Day 210 and Day 365
Frequencies of HPV-16 and -18 specific B-cells measured by B-cell ELISPOT | Day 0, Day 45, Day 180, Day 210 and Day 365
B-cell profile measured by Flow cytometry | Day 0, Day 45, Day 180, Day 210 and Day 365
Secretion of pro- and antiinflammatory cytokines from PBMC's stimulated with innate stimuli measured by Luminex or Elisa | Day 0, Day 45, Day 180, Day 210 and Day 365
Type-specific HPV-DNA from cervical and genital swab material | Day 0 and Day 210
CD4 cell count and HIV viral load | Day 0, Day 45, Day 180, Day 210 and Day 365
Occurrence and intensity of solicited local symptoms | Day 0-6 after each vaccination
  Participants will complete a vaccination diary with regards to local symptoms. Number and intensity of local symptoms will be listed and summarized.
Occurrence, intensity and relationship to vaccination of solicited general symptoms | Day 0-6 after each vaccination
  Participants will complete a vaccination diary with regards to general symptoms. Number and intensity of generalized symptoms will be listed and summarized in a form.
Occurrence of SAEs | Throughout the active phase of the study (up to Day 210)
Occurrence of clinically relevant abnormalities in hematological and biochemical parameters | Throughout the active phase of the study (up to Day 210)
  Clinical significant changes in hemoglobin, ALAT, basic phosphatase and creatinine compared to baseline values will be listed and summarized.
Geometric mean titres of HPV-16 and HPV-18 and total Immunoglobulin G (IgG) titers in cervicovaginal secretion (CVS) from female participants | Day 0, Day 210 and Day 365
Geometric mean titres of serum HPV-6 and HPV-11 antibody measured by a competitive Luminex immunoassay (cLIA) | To be measured at day 0, day 45, day 180, day 210 and day 365
% of participants seropositive for anti-HPV-6, -11 -18, -31, -33, -45, -52 and -58 | Day 0, Day 45, Day 180, Day 210, Day 365
  % of participants seropositive for anti-HPV-6, -11 as measured by a competitive Luminex immunoassay (cLIA) and % of participants seropositive for anti-HPV-18, -31, -33, -45, -52 and -58 antibodies as measured by either Pseudovirion-Based Neutralization Assay (PBNA)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Østergaard, MD,PhD,DmSC, Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark; Lars Toft, MD, Principal Investigator — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Toft L, Tolstrup M, Muller M, Sehr P, Bonde J, Storgaard M, Ostergaard L, Sogaard OS. Comparison of the immunogenicity of Cervarix(R) and Gardasil(R) human papillomavirus vaccines for oncogenic non-vaccine serotypes HPV-31, HPV-33, and HPV-45 in HIV-infected adults. Hum Vaccin Immunother. 2014;10(5):1147-54. doi: 10.4161/hv.27925. Epub 2014 Feb 19. PMID 24553190
- [Derived] Toft L, Storgaard M, Muller M, Sehr P, Bonde J, Tolstrup M, Ostergaard L, Sogaard OS. Comparison of the immunogenicity and reactogenicity of Cervarix and Gardasil human papillomavirus vaccines in HIV-infected adults: a randomized, double-blind clinical trial. J Infect Dis. 2014 Apr 15;209(8):1165-73. doi: 10.1093/infdis/jit657. Epub 2013 Nov 23. PMID 24273179